CLINICAL TRIAL: NCT04988581
Title: Effectiveness of Intensively Integrated Care of Microvascular Risk Factors to Prevent Diabetic Kidney Disease Incidences in Community Clinics in Xiamen, China: An Open-label Randomized Controlled Trial
Brief Title: Prevention In Community Clinics From Diabetic Kidney Disease
Acronym: PICK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KYH2021-032
Record Dates: First submitted 2021-07-13; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Diabetic Nephropathies
Keywords: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensively Integrated Care of Microvascular Risk Factors (Experimental): intensively integrated care of microvascular risk factors (glycated hemoglobin [HbA1C], urinary albumin-to-creatinine ratio [ACR], blood pressure [BP], estimated glomerular filtration rate [eGFR], uric acid [UA] and low-density lipoprotein cholesterol [LDL])
  Interventions: Other: Intensively integrated care of microvascular risk factors in the intervention group
- Usual Care of Microvascular Risk Factors (No Intervention): Usual care among patients with diabetes

INTERVENTIONS:
Other: Intensively integrated care of microvascular risk factors in the intervention group — The intensively integrated care, which will provide a standardized, combined, multi-component intervention according to clinical guideline treatment for diabetes and comorbidities in a primary care setting, will be delivered by trained primary care physicians, health managers and diabetes specialists. Diabetic microvascular risk factors (glycated hemoglobin [HbA1C], urinary albumin-to-creatinine ratio [ACR], blood pressure [BP], estimated glomerular filtration rate [eGFR], uric acid [UA] and low-density lipoprotein cholesterol [LDL]) will be tested every 3 month for the intervention group and clinical treatment decisions based on the test results will be implemented accordingly when necessary. The intensively integrated care intervention will last for 36 months. HbA1C, ACR, BP, eGFR, UA, LDL, other variables and co-morbidities will be measured at baseline and follow-up visits every 3 month.
  Arms: Intensively Integrated Care of Microvascular Risk Factors

SUMMARY:
The overall objective of the proposed randomized trial is to test whether implementation of intensively integrated care of microvascular risk factors (glycated hemoglobin [HbA1C], urinary albumin-to-creatinine ratio [ACR], blood pressure [BP], estimated glomerular filtration rate [eGFR], uric acid [UA] and low-density lipoprotein cholesterol [LDL]) will improve and reduce diabetic kidney disease events (DKD morbidity and mortality) among patients with diabetes and additional microvascular risk factors compared to usual care in public primary care setting (community health service center) in Xiamen, China.

DETAILED DESCRIPTION:
Most patients with diabetes, which has reached epidemic proportions in China, have multiple uncontrolled microvascular risk factors due to suboptimal care. Diabetic kidney disease events (DKD) is one of the most common microvascular complications and has been becoming the leading cause of end-stage renal disease (ESRD).

The overall objective of the proposed randomized trial is to test whether implementation of intensively integrated care of microvascular risk factors (glycated hemoglobin [HbA1C], urinary albumin-to-creatinine ratio [ACR], blood pressure [BP], estimated glomerular filtration rate [eGFR], uric acid [UA] and low-density lipoprotein cholesterol [LDL]) will improve and reduce diabetic kidney disease events (DKD morbidity and mortality) among patients with diabetes and additional microvascular risk factors compared to usual care in public primary care setting (community health service center) in Xiamen, China.

The Prevention In Community Clinics From Diabetic Kidney Disease (PICK) study is an open-label randomized controlled trial which will be conducted in one public primary care setting (Lianqian community health service center) in Xiamen, China. The proposed trial will recruit 1240 patients with diabetes and additional microvascular risk factors but without DKD at baseline. Approximately 620 participants will be randomly assigned to the intervention group and similar participants to the control group.

The intensively integrated care, which will provide a standardized, combined, multi-component intervention according to clinical guideline treatment for diabetes and comorbidities in a primary care setting, will be delivered by trained primary care physicians, health managers and diabetes specialists. Diabetic microvascular risk factors (glycated hemoglobin [HbA1C], urinary albumin-to-creatinine ratio [ACR], blood pressure [BP], estimated glomerular filtration rate [eGFR], uric acid [UA] and low-density lipoprotein cholesterol [LDL]) will be tested every 3 month for the intervention group and clinical treatment decisions based on the test results will be implemented accordingly when necessary. The intensively integrated care intervention will last for 36 months. HbA1C, ACR, BP, eGFR, UA, LDL, other variables and co-morbidities will be measured at baseline and follow-up visits every 3 month. Meanwhile management of the diabetic microvascular risk factors for the control group will be conducted as usual.

In Phase 1, the primary outcomes are mean reductions in HbA1C, ACR, BP, eGFR, UA and LDL levels over the 18-month intervention between intervention and control groups. Net change in HbA1C, ACR, BP, eGFR, UA and LDL levels will be simultaneously modeled using a scaled marginal model which allows estimation of a single overall intervention effect.

In Phase 2, the primary outcome is differences in DKD morbidity and mortality over the 36-month intervention between intervention and control groups.

The secondary outcomes are the cumulative incidence rates of albuminuria and renal impairment over 36-months of intervention.

The proposed trial is designed to provide 80% statistical power to detect a 4% reduction in the cumulative incidence of DKD at a 2-sided significance level of 0.05. An 90% follow-up rate is assumed and is taken into consideration in the power calculation.

This implementation research project has a high impact in public health, because it will generate urgently needed data on an effective, practical, and sustainable intervention program aimed at reducing DKD burden among diabetes patients in developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes patients
* Men or women aged 30-75 years who received primary care from the Lianqian clinics in Xiamen, China
* Patients with at least one microvascular risk factors (glycated hemoglobin [HbA1C], urinary albumin-to-creatinine ratio [ACR], blood pressure [BP], estimated glomerular filtration rate [eGFR], uric acid [UA] and low-density lipoprotein cholesterol [LDL]) .

Exclusion Criteria:

* Diabetic Kidney Disease
* Patients with heart failure, or receiving hemodialysis, or with contraindications to metformin or statin treatments
* Women who are pregnant or plan to become pregnant
* Patients who cannot be followed for 36 months
* Patients who are unwilling or unable to give informed consent

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1240 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1 | 18 months
  In Phase 1, the primary outcomes are mean changes in HbA1C, ACR, BP, eGFR, UA and LDL levels over the 18-month intervention between intervention and control groups.
Phase 2 | 36 months
  In Phase 2, the primary outcome is differences in DKD morbidity and mortality over the 36-month intervention between intervention and control groups.

SECONDARY OUTCOMES:
The secondary outcomes | 36 months
  The secondary outcomes are the cumulative incidence rates of albuminuria and renal impairment over the 36-month individually over 36-months of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Zhibin Li, Ph.D., Principal Investigator — The First Affiliated Hospital of Xiamen University